CLINICAL TRIAL: NCT05793086
Title: Electrophysiological and Ultrasound Quantitative Biomarkers for Myofascial Pain
Brief Title: Evaluation of a Novel Class of Objective Myofascial Pain Assessments
Acronym: ENCOMPASS
Status: Active, not recruiting | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Seward Rutkove, Neurology Department Chair, Beth Israel Deaconess Medical Center
Other Study IDs: 2022P000543
Record Dates: First submitted 2023-03-19; First posted 2023-03-31 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Myofascial Pain; Trigger Point Pain, Myofascial
Keywords: Myofascial Pain; Trigger point
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (3):
- active trigger point group: Individuals with active trigger points in trapezius
  Interventions: Diagnostic Test: Ultrasound; Diagnostic Test: Electrical impedance myography; Diagnostic Test: Excitability testing
- latent trigger point group: Individuals with trigger points in trapezius without spontaneous pain
  Interventions: Diagnostic Test: Ultrasound; Diagnostic Test: Electrical impedance myography; Diagnostic Test: Excitability testing
- healthy trapezius muscle: Individuals without trigger points.
  Interventions: Diagnostic Test: Ultrasound; Diagnostic Test: Electrical impedance myography; Diagnostic Test: Excitability testing

INTERVENTIONS:
Diagnostic Test: Ultrasound — Using shear wave elastography and gray scale analysis of ultrasound.
Diagnostic Test: Electrical impedance myography — Measurement of localized bioimpedance of muscle
Diagnostic Test: Excitability testing — Electrical studies of myofiber excitability

SUMMARY:
This is an observational study that is intended to determine the capacity of three technologies to serve as diagnostic biomarkers for myofascial pain syndrome. Investigators will seek patients with myofasical pain syndrome as well as healthy subjects for this study. Electrical impedance myography (EIM), myofiber threshold tracking (TT) excitability testing, and ultrasound with shear wave elastography (SWE) measurements will be obtained from the trapezius muscle (the muscle that extends over the back of the neck and shoulders). These measurements will be repeated within 2-5 days to assess repeatability of these methods.

DETAILED DESCRIPTION:
Study Visit One:

1. Overview
2. History and examination (All participants). After reviewing the purpose and procedures of the study, the subject, or a legally authorized representative (LAR), will be asked to sign the internal review board-approved informed consent form.

   Basic medical, social, and family histories will then be obtained and recorded. Previous medical records will be reviewed. Medications, including drug doses, history of recent medication changes, and duration of treatment) will be reviewed.

   A brief physical exam will be performed. If the subject has MPS, the study doctor will identify the trigger points and will mark those with a permanent marker.
3. Electrical Impedance Myography (EIM) - a trained technician will apply several small sticky pads (electrodes) to different parts of the subject's muscle and a very tiny electrical current will be applied that they will not feel. Several measurements will be done their muscle. This will take approximately 10 minutes
4. Ultrasound (US) - a trained technician will apply a small amount of gel to the skin. They will hold a small hand-held device on the skin and will measure the muscle. The gel is easily cleaned off of the skin when the testing is complete. This will take approximately 20 minutes
5. Threshold Tracking (TT) - TT tests how quickly muscle responds to stimulation. The muscle is stimulated using a small needle which is placed superficially in their trapezius muscle. The subject will feel a small needle prick which should be less uncomfortable than having blood drawn. Electrodes (small sticky pads) are placed a short distance from the needle over the muscle. When their muscle is stimulated with the needle, the time it takes for the muscle to react is measured by the electrodes. This procedure will last 30 minutes and creates a tingling feeling.
6. Questionnaires- Subjects will be asked to complete some brief questionnaires about their pain, mood, and sleep. Overall, this visit will take approximately 1 - 1.5 hours.

Home Period Subjects will be asked to re-inforce/re-apply the permanent marker spots made at their first visit. This is so investigators can use the same spots for testing at the next visit.

Study Visit 2 (2-14 days after Study Visit #1) The second study visit is identical to the first one. A study team member will test the subject's trigger points again at the beginning of the visit. This visit will also last approximately 1-1.5 hours.

ELIGIBILITY:
Myofascial Pain Syndrome with active and/or latent TrPs

Inclusion Criteria:

1. Ages: 18-80
2. Myofascial Pain Syndrome with active and/or latent TrPs, as diagnosed by a pain specialist, with involvement of the trapezius meeting criteria (detailed in "Methods"))
3. Capacity to manage breakthrough pain medications during the study with only acetaminophen

Exclusion Criteria:

1. Presence of radicular pain, superimposed neuromuscular disease, or condition
2. Fibromyalgia or other generalized pain condition
3. Opioid use
4. Active mood or substance use disorder
5. Taking or unable to wean off pain medications that directly affect neuronal or muscle excitability at least 2 weeks prior to study enrollment and remain off for the duration of the study: gabapentin, pregabalin, topiramate, carbamazepine, oxcarbazepine, valproic acid, tricyclic antidepressants (such as nortriptyline and amitriptyline), tizanidine, cyclobenzaprine, carisoprodol, methocarbamol, benzodiazepines
6. Skin allergy or sensitivity that would preclude the use of adhesive electrodes
7. Systemic or psychiatric illness that in the opinion of the Site Investigator would interfere with the individual's ability to participate in the trial.
8. Anticoagulation (with coumadin, clopidogrel, or direct oral anticoagulants; aspirin acceptable).

Healthy volunteers

Inclusion Criteria:

1. Ages: 18-80

Exclusion Criteria:

1. Presence of radicular, myofascial, or generalized pain, superimposed neuromuscular disease or condition
2. History of MPS, examination demonstrating trigger points
3. Fibromyalgia or other generalized pain condition
4. Opioid use
5. Active mood or substance use disorder
6. Taking or unable to wean off pain medications that directly affect neuronal or muscle excitability at least 2 weeks prior to study enrollment and remain off for the duration of the study: gabapentin, pregabalin, topiramate, carbamazepine, oxcarbazepine, valproic acid, tricyclic antidepressants (such as nortriptyline and amitriptyline), tizanidine, cyclobenzaprine, carisoprodol, methocarbamol, benzodiazepines
7. Skin allergy or sensitivity that would preclude85 the use of adhesive electrodes
8. Systemic or psychiatric illness that in the opinion of the Site Investigator would interfere with the individual's ability to participate in the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with myofascial pain syndrome with active and/or latent TrPs, as diagnosed by a pain specialist, with involvement of the trapezius meeting
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-01-27 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Primary outcome: Electrical Impedance Myography (EIM) | 2.5 years
  The primary outcome will be 100 kHz phase angle in EIM

SECONDARY OUTCOMES:
Secondary outcome: Ultrasound with shear wave elastography (SWE) | 2.5 years
  echointensity and elastic modulus
Secondary outcome: Excitability threshold tracking (TT) | 2.5 years
  The secondary outcome will be maximum latency change with a conditioning stimulus

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
When the project is finished and all primary analyses are complete, a final, complete, cleaned, and de-identified data set will be provided for public access including the appropriate data dictionaries and case report forms. In addition to the sharing of resources during the trial, the investigators of this study are fully committed to participate in data sharing as per NIH policies. Following completion of all planned analyses and manuscripts, investigators will make the data and associated documentation available to qualified users though repositories like the Biomedical Informatics Research Network (BIRN), which is capable of supporting large volumes of data (e.g. neuroimaging), and NIH HEAL Initiative Central Data Repository.